Official Title: Dietary behaviour change intervention on managing sarcopenic obesity in community-dwelling older people: a feasibility and pilot study

Date of the document: 19/10/2020

Approved by the Human Subjects Ethics Sub-committee of The Hong Kong Polytechnic University on 15/10/2019



## CONSENT TO PARTICIPATE IN RESEARCH

## Dietary behaviour change intervention on managing sarcopenic obesity in community-dwelling older people: a feasibility and pilot study

Principal Investigator: Dr. Justina Yat Wa LIU, Co-Principal Investigator: Prof. Maritta VÄLIMÄKI, Ms Yueheng YIN hereby consent to participate in the captioned research conducted by Justina Yat Wa LIU. I understand that information obtained from this research may be used in future research and published. However, my right to privacy will be retained, i.e. my personal details will not be revealed. The procedure as set out in the attached information sheet has been fully explained. I understand the benefit and risks involved. My participation in the project is voluntary. I acknowledge that I have the right to question any part of the procedure and can withdraw at any time without penalty of any kind. **Participant:** Name of Participant Signature Date Researcher: Name of Researcher Signature Date



## **INFORMATION SHEET**

## Dietary behaviour change intervention on managing sarcopenic obesity in communitydwelling older people: a feasibility and pilot study

Principal Investigator: Dr. Justina Yat Wa LIU, Co-Principal Investigator: Prof. Maritta VÄLIMÄKI, Ms Yueheng YIN

You are invited to participate in this research project. The project has been approved by the Human Subjects Ethics Sub-committee (HSESC) (or its Delegate) of The Hong Kong Polytechnic University (HSESC Reference Number: 20191007001). The aims of this project are to examine the feasibility and the preliminary effects of the dietary behaviour change intervention on body composition for older people with sarcopenic obesity.

If you decide to be in this study, your socio-demographic data will be obtained for research and education purpose. Each participant will be randomized to either the dietary intervention group or the control group. The dietary intervention group will receive a 15-week dietary behavior change intervention tailored with 6 face-to-face meetings and weekly telephone call. The control group will not be required to do anything, the participants will only receive regular social contacts with similar frequency as the dietary intervention group.

To further understand the acceptability of the dietary intervention, 10 to 15 participants from the dietary intervention group will be invited to attend individual semi-structured interview. Your response to interview questions will be kept confidential.

Adverse events such as hypoglycemia or anorexia may arise during the dietary intervention process. Therefore, the potential adverse events relating to the intervention will be discussed with you. All information related to you will remain confidential and will be identifiable by codes only known to the researchers. The collected data may be used for future studies, education and academic purposes.

You have every right to withdraw from the study before or during the measurement without penalty of any kind. If you have any questions, you may ask our helpers now or later, even after the study has started.

You may contact Dr Justina Liu at (852) 2766 4097.

If you have any complaints about the conduct of this research study, you may contact the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University in writing (c/o Research Office of the University) stating clearly the responsible person and department of this study as well as the HSESC Reference Number.

Thank you for your interest in participating in this study.

Dr. Justina Yat Wa LIU Principal Investigator